CLINICAL TRIAL: NCT01412437
Title: Multimodal Neuroimaging and Neurocognitive Assessment of Biomarkers and Response to Sapropterin Dihydrochloride Treatment in Phenylketonuria
Brief Title: Neuroimaging and Neurocognitive Assessment and Response to Sapropterin Dihydrochloride Treatment in Phenylketonuria
Acronym: PKU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Children's National Research Institute (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Andrea Gropman, Associate Professor, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BMRN 9956
Record Dates: First submitted 2011-08-01; First posted 2011-08-09 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: PKU
Keywords: PKU; MRI; neurocognition; sapropterin dihydrochloride
MeSH Terms: interventions — Diet; sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet (Experimental): 12 participants will be randomized to diet. Phe levels will be followed by blood levels. A dietician will analyze diet for phe content and advise
  Interventions: Dietary Supplement: diet
- sapropterin dihydrochloride (Experimental): Intervention: 24 participants will be randomized to receive the drug 10 mg/kg per day. Responders and non responders will remain on drug for four months
  Interventions: Drug: sapropterin dihydrochloride

INTERVENTIONS:
Dietary Supplement: diet — 12 participants will be randomized to diet. Phe levels will be followed by blood levels. A dietician will analyze diet for phe content and advise
  Other Names: PKU diet
  Arms: Diet
Drug: sapropterin dihydrochloride — 20 mg/kg for 4 months
  Other Names: Biomarin Kuvan
  Arms: sapropterin dihydrochloride
Drug: sapropterin dihydrochloride
  Other Names: Kuvan
  Arms: sapropterin dihydrochloride

SUMMARY:
The investigators will use different types of brain imaging (MRI) in patients with Phenylketonuria (PKU) who are currently not on a strict diet to test the hypothesis that there is improvement in brain circuitry and biochemistry after return to diet and/or sapropterin dihydrochloride (Kuvan).

DETAILED DESCRIPTION:
We plan to enroll 36 subjects with PKU. They will all be counseled to follow the PKU diet. They will be randomized to receive Kuvan. We will plan to enroll 12 in the diet alone group and 24 in the Kuvan group with the hope of 12 being responders (as defined by a 30% drop in blood phe levels). Those who do not have a blood response with decreased Phe will still be evaluated for a neurological response as measured by neurocognitive testing and neuroimaging as outlined in this protocol. All 24 in the Kuvan group will receive a 1 month trial of Kuvan and then the responders will have their insurance cover the drug and for the non responders Biomarin will supply Kuvan.

Aim 1: To test the hypothesis that stable patients with PKU who are not currently on diet have specific brain biomarkers quantifiable by DTI, fMRI and MRS and that the levels of these biomarkers correlate with the clinical severity and outcome. Our pilot study and the research of others have suggested the following as potential biomarkers for neural injury in PKU:

* Metabolic abnormalities: elevated Phe concentrations as measured by MRS.
* White matter microstructure: measured by apparent diffusion coefficient, (ADC), using DTI.
* Working memory and attention/executive function: measured by fMRI, Near infrared spectroscopy (NIRS) and neuropsychological testing.

We will study these potential biomarkers in a group of well characterized adults with PKU who are not currently on diet or a strict diet as evidenced by elevated Phe, but who were identified by the newborn screen and may have been on diet during childhood, with varying severity of clinical involvement.

Aim 2: To measure changes in biomarkers validated in Aim 1 after return to diet +/- Kuvan (sapropterin dihydrochloride; Kuvan)

Based on our preliminary data and that of others, Aim 1 should provide us with a number of candidate biomarkers for brain injury in PKU. We expect that these will include three types of markers that can be correlated: metabolic, structural and cognitive. We will use these biomarkers to study subjects during return to diet and/or initiation of Kuvan.

Aim 3: To compare cognitive performance in our subjects prior to and after return to diet +/- Kuvan. using the following tests:

Comprehensive Trail making test (CTMT) -Parts A and B Stroop WASI (IQ, digit span) BRIEF Edinburgh Handedness Inventory Hand Preference Demonstration Test

Outcome variables The primary endpoints in this study are 1) an estimate of the white matter damage (macroscopic and microscopic) in participants with PKU versus controls at baseline and after return to diet +/- Kuvan; 2) determination of a profile of brain biochemical abnormalities in participants with PKU versus controls at baseline and after return to diet/Kuvan, 3) assessment of cognitive and motor systems abnormalities (by fMRI and cognitive testing) in the participant cohort as compared to age matched typically developing non disease controls at baseline and after return to diet/Kuvan; 4) coefficient of variability of scoring on traditional neurocognitive.

After the conclusion of this study, future areas of research would include expansion to study long term effects of Kuvan, study of more impaired populations and response to Kuvan, and using optical imaging methods we are currently piloting in OTCD.

Method to investigate biomarkers of disease We plan to use 1HMRS to identify markers of disease severity such as elevations of Phe and decreases in NAA. This will be compared in participants and normal age matched controls. Additionally, diffusion tensor imaging will allow us to probe white matter fiber tracts that may be especially vulnerable in this disorder selectively. Lastly, fMRI may identify regions of differential activation in the brain that are different in participants versus age matched controls at rest and with a cognitive task probing working memory and attention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PKU identified on Newborn screening and with phe concentration >12mg/dl on the newborn screen
2. Baseline phe level at study enrollment > 20 mg/dl (this is the level required for inclusion in the study, regardless of the level used to make diagnosis)
3. Age range: 18-45 years
4. Able to comply with neuroimaging without requiring sedation (typically requires IQ over 65). The IQ will be checked with the WASI (Weschler Adult scales of intelligence) before determining eligibility
5. Able to undergo neuroimaging safely (i.e. without presence of ferromagnetic devices)
6. Subject has ability to follow instructions in English
7. Female of childbearing age who is sexually active agrees to urine pregnancy test
8. Availability to come to Washington, DC to participate in this study

Exclusion Criteria:

1. Age range <18 or >45 years
2. Inability to comply with neuroimaging without the use of sedation (low IQ or claustrophobic)
3. Presence of ferromagnetic device(s) that preclude safe imaging including cardiac pacemaker, neural pacemaker, surgical clips in the brain or blood vessels, surgically implanted metal plates, screws or pins, cochlear implants or metal objects in their body
4. Pregnant female or breastfeeding at screening or planning to become pregnant at any time during the study.
5. Baseline phe < 20 mg/dl
6. Currently on Kuvan
7. History of substance abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Neuroimaging biomarkers | at 4 months
  An estimate of the change in white matter damage and biochemistry in participants with PKU after either diet/Kuvan

SECONDARY OUTCOMES:
Brain biochemistry | at 4 months
  Assessment of cognitive systems abnormalities (by fMRI ) in the participant cohort after diet/Kuvan

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Gropman, M.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Christ SE, Moffitt AJ, Peck D. Disruption of prefrontal function and connectivity in individuals with phenylketonuria. Mol Genet Metab. 2010;99 Suppl 1:S33-40. doi: 10.1016/j.ymgme.2009.09.014. PMID 20123468